CLINICAL TRIAL: NCT07267494
Title: Image-guided Herniorrhaphy Safety and Efficacy Pilot
Brief Title: Image-Guided Herniorrhaphy Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2345685
Record Dates: First submitted 2025-11-10; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hernia; Hernia Abdominal Wall; Ventral Hernia; Inguinal Hernia; Hiatal Hernia; Diastasis Recti
Keywords: Image-guided herniorrhaphy; hernia; pilot study; quality of life; safety and feasability
MeSH Terms: conditions — Hernia; Hernia, Abdominal; Hernia, Ventral; Hernia, Inguinal; Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: All participants will undergo a single, image-guided, needle-based herniorrhaphy procedure performed under ultrasound and/or CT guidance with local anesthesia and optional sedation. This pilot is designed to assess procedural safety and changes in hernia-related quality of life to determine feasibility for a larger trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image-Guided Herniorrhaphy (Experimental): Single-arm pilot. All participants undergo a percutaneous, image-guided needle-based hernia repair performed under ultrasound and/or CT guidance with local anesthesia and optional moderate sedation. Follow-up includes clinic visits and quality-of-life assessments over ~8 months.
  Interventions: Procedure: Image-Guided Herniorrhaphy

INTERVENTIONS:
Procedure: Image-Guided Herniorrhaphy — Minimally invasive, image-guided repair of abdominal or groin hernias. Under ultrasound (primary) and, when indicated, low-dose CT guidance, a hollow needle preloaded with bi-directional barbed suture is passed percutaneously across the defect to approximate and secure tissue without surgical incisions or general anesthesia. The procedure is performed in the interventional radiology suite with local anesthesia and optional moderate IV sedation; typical procedure time ~30-60 minutes. Standard post-procedure monitoring is completed prior to discharge.
  Arm/Intervention Link: Applied to the "Image-Guided Herniorrhaphy" (Experimental) arm.

SUMMARY:
This pilot clinical study will evaluate the safety and effectiveness of a new image-guided, needle-based approach for repairing abdominal or groin hernias in adults who are unable or unwilling to undergo traditional open or laparoscopic surgery. The technique uses ultrasound and, when needed, CT imaging to guide a hollow needle preloaded with barbed suture through the skin to close the hernia defect without large incisions or general anesthesia. Each participant will undergo one image-guided procedure and will be followed for eight months to assess complications and changes in hernia-related quality of life. Approximately thirty participants will be enrolled. The study aims to determine whether this minimally invasive approach is safe, feasible, and capable of improving hernia symptoms enough to justify a larger clinical trial

DETAILED DESCRIPTION:
Traditional hernia repair requires either open surgical incisions or laparoscopic entry into the abdomen, typically under general anesthesia. Although effective, these operations can be unsuitable for frail or medically complex patients because of anesthesia risks, postoperative pain, and wound complications.

This investigator-initiated pilot study explores a minimally invasive alternative: a percutaneous, image-guided herniorrhaphy that uses ultrasound or CT to visualize the hernia and guide placement of a barbed suture through a hollow needle to close the tissue defect. The goal is to assess procedural safety, feasibility, and short-term improvement in hernia-related quality of life.

Participants will be adults with reducible abdominal, groin, or hiatal hernias who are not candidates for standard surgery. The study procedure will be performed in the interventional radiology suite using local anesthesia with or without moderate sedation, following existing institutional workflows for other needle-based image-guided procedures.

Safety monitoring is provided by two independent physicians-a hernia surgeon and an interventional radiologist-who review study data quarterly and have authority to pause or stop the study if predefined complication criteria are met. Safety events will be categorized using the Society of Interventional Radiology adverse-event classification.

This study is intended to generate preliminary data on safety and patient-reported outcomes that can inform future trials of image-guided hernia repair techniques.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult with reducible hernia(s) or diastasis smaller than approximately 8 cm seeking treatment for their hernia but not able or willing to undergo traditional surgery (open, laparoscopic, or robotic)
* Patient must be willing to undergo a novel 30- to 60-minute image-guided needle-based procedure

Exclusion Criteria:

* Children, prisoners, and pregnant women (possibly requiring a pregnancy test on the day of the procedure)
* Patients with a known reaction to local anesthetic or sedation medications or the suture material to be used
* Patients with irreducible hernias
* Patients with herniation not visible by ultrasound or CT
* Patients that do not fit the diameter of a CT gantry or the weight limit of the procedural CT table
* Patients without insurance or not willing to pay out-of-pocket for the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the Image-Guided Herniorrhaphy Procedure | Through 8 months after the procedure
  Frequency, type, and severity of all procedure-related adverse events, categorized according to the Society of Interventional Radiology (SIR) Adverse Event Classification. Major complications (e.g., bleeding, bowel injury, infection, or events requiring hospitalization >48 hours) and minor complications will be recorded and reviewed by independent safety monitors.
Change in Hernia-Related Quality of Life (Short Form-36 Health Survey) | Through 8 months after the procedure
  Mean change in general health-related quality-of-life scores measured using the Short Form-36 (SF-36) Health Survey, a validated 36-item measure assessing eight domains of physical and mental health. Scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in Hernia-Specific Quality of Life (Hernia-Related Quality-of-Life Survey) | Through 8 months after the procedure
  Mean change in hernia-specific quality-of-life scores measured using the Hernia-Related Quality-of-Life Survey (HerQLes), a validated 12-item instrument used for ventral and abdominal wall hernias. Scores range from 0 to 100, with higher scores indicating better hernia-related quality of life.
Change in Reflux-Related Quality of Life (GERD-Health-Related Quality of Life Questionnaire) | Through 8 months after the procedure
  Mean change in symptom severity and quality-of-life scores measured using the Gastroesophageal Reflux Disease-Health-Related Quality of Life (GERD-HRQL) questionnaire, a validated 10-item scale used in patients with hiatal hernias. Scores range from 0 to 75, with higher scores indicating worse reflux symptoms and lower quality of life.

SECONDARY OUTCOMES:
Incidence of Delayed Adhesion-Related Symptoms | Up to 8 months after procedure
  Number of participants reporting new or worsening abdominal pain, nausea, vomiting, or bowel obstruction potentially related to intra-abdominal adhesions, assessed via follow-up visits and phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larson, MD, Principal Investigator — UC Davis Health - Department of Radiology
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No